CLINICAL TRIAL: NCT06020989
Title: A Randomized, Phase 2 Trial of Lazertinib and Chemotherapy Combination in EGFR-mutant NSCLC Patients Without ctDNA Clearance After lead-in Lazertinib Monotherapy (CHAMELEON)
Brief Title: Lazertinib and Chemotherapy Combination in EGFR-mutant NSCLC Patients Without ctDNA Clearance After lead-in Lazertinib Monotherapy
Acronym: CHAMELEON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0795
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Lazertinib + chemotherapy combination
  Interventions: Drug: Lazertinib+Pemetrexed+Carboplatin
- B (Active Comparator): Lazertinib monotherapy
  Interventions: Drug: Lazertinib
- C (Active Comparator): Lazertinib monotherapy
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib+Pemetrexed+Carboplatin — Arm A will receive Lazertinib and Pemetrexed, Carboplatin combination. Lazertinib will be given 240 mg once a day daily PO until disease progression or unacceptable toxicity. Pemetrexed(500 mg/m2) will be administered IV infusion on Day 1 of each 21-day cycle until disease progression or unacceptable toxicity. Carboplatin(AUC5) will be administered IV infusions on Day 1 of each 21-day cycle until 4 cycles.
  Arms: A
Drug: Lazertinib — Lazertinib will be given 240 mg once a day daily PO until disease progression or unacceptable toxicity.
  Arms: B
Drug: Lazertinib — Lazertinib will be given 240 mg once a day daily PO until disease progression or unacceptable toxicity.
  Arms: C

SUMMARY:
Lazertinib is an oral third-generation irreversible tyrosine kinase inhibitor (TKI) that has proved to selectively inhibit EGFR-TKI sensitizing mutations (exon 19 deletion or exon 21 L858R) and be effective in patients with central nervous system (CNS) metastases. However, all patients eventually experience disease progression. For patients with MRD, lazertinib plus cytotoxic anticancer drug can prolong the duration of response or even induce complete cure, indicating this combined treatment strategy is considered the safest and most effective.

The objective of this phase 2 prospective two-arm clinical trial is to evaluate the safety and efficacy of lazertinib alone or in combination with cytotoxic chemotherapy in EGFR-mutant (exon 19 deletion or exon 21 L858R) NSCLC patients without ctDNA clearance after lead-in lazertinib. If anticancer drugs are used only for patients with MRD, the risk of resistance development will decrease, improving PFS.

Hypothesis: to evaluate the efficacy defined as the PFS rate of lazertinib alone or in combination with a cytotoxic anticancer drug in EGFR-mutant NSCLC patients without ctDNA clearance after lead-in lazertinib monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed recurrent or metastatic non-squamous NSCLC without previous treatment experience
2. Presence of the sensitising EGFR-mutation (exon 19 deletion and/or L858R) detected by an accredited laboratory.
3. Measurable disease as defined according to RECIST v1.1
4. Age ≥19 years
5. ECOG performance status 0-2
6. Life expectancy ≥12 months
7. Adequate haematological function:

   1. Haemoglobin ≥90 g/L
   2. Absolute neutrophil count (ANC) ≥ 1.5× 109/L
   3. Platelet count ≥100× 109/L
8. Adequate renal function:

   1. Serum creatinine ≤1.5x ULN or creatinine clearance ≥50 mL/min (calculated according to Cockcroft-Gault formula, see below).
   2. Confirmation of creating clearance is only required when serum creatinine is >1.5x ULN.

   Cockcroft-Gault formula:"mL" /"min" "=" ("140-age" ["years" ])"×actual body weight " ["kg" ]/("72×" 〖"Creatinine" 〗_"serum" " " ("mg" /"dL" ) ) "(×0.85 if female)"
9. Adequate liver function:

   1. ALT and AST ≤2.5× ULN. If the patient has liver metastases, ALT and AST must be ≤5× ULN
   2. Total serum bilirubin ≤1.5× ULN. If the patient has documented Gilbert's syndrome (unconjugated hyperbilirubinaemia) ≤3× ULN.
10. Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 7 days before enrolment.
11. Written IC for protocol treatment must be signed and dated by the patient and the investigator prior to any trial-related intervention.

Exclusion Criteria:

1. Presence of leptomeningeal metastases
2. Symptomatic spinal cord compression
3. Currently receiving (or unable to stop use prior to receiving the first dose of lazertinib treatment) medications or herbal supplements known to be potent CYP3A4 inducers that cannot be stopped before enrolment and for the duration of the trial.
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
5. Patients with a resolved or chronic HBV infection are eligible if they are:

   1. Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG]; or
   2. Positive for HBsAg, negative for HBeAg but for >6 months have had transaminases levels below ULN and HBV DNA levels below 2000 IU/mL (i.e., are in an inactive carrier state).
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of lazertinib
7. Any of the following cardiac criteria:

   1. QTcF >470 msec obtained from 3 ECGs, using the screening clinic ECG machine derived QTc value (QTcF: corrected QT interval using Fridericia's formula).
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block or second-degree heart block).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes (TdP).
8. Past medical history of ILD, drug induced ILD, interstitial pneumonitis which required steroid treatment, or any evidence of clinically active ILD
9. History of hypersensitivity to active or inactive excipients of lazertinib or drugs with a similar chemical structure or class to lazertinib.
10. Patients who should not participate in the trial at the investigator's discretion as they are unlikely to comply with trial procedures, restrictions, and requirements for pregnant or lactation women.
11. Both sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method (Please refer to 8.3 for highly effective contraceptive methods) during the trial and up to 6 months after discontinuing lazertinib treatment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS is measured from the date of start of study to the date of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Min Lim, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No